CLINICAL TRIAL: NCT04516590
Title: The Diagnostic Value of Autoimmune Antibody Detection in Newly Onset and Chronic Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: General Hospital of Ningxia Medical University (Other); LanZhou University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Henan Provincial People's Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); Wulumuqi General Hospital of Lanzhou Military Command (Other); Xuanwu Hospital, Beijing (Other); Xiangya Hospital of Central South University (Other); West China Hospital (Other); Affiliated Hospital of Qinghai University (Other)
Responsible Party: Sponsor
Other Study IDs: XijingH Deng Yanchun-1
Record Dates: First submitted 2020-06-30; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Epilepsy
Keywords: epilepsy; autoimmune antibody; diagnose
MeSH Terms: conditions — Epilepsy; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- autoimmune antigen negative: treated with anti-epilepsy drugs
- autoimmune antigen positive: whether the patients receive immune therapy or not will depend on the type and titter of the autoimmune antibody as well as the severity of the symptom

INTERVENTIONS:
Other:  — There was no intervention in this observational study

SUMMARY:
multi-central and prospectively study the diagnostic value of autoimmune antibody detection in new and chronic epilepsy, and provide reference for clinical practice

DETAILED DESCRIPTION:
multi-centrally recruit patients with newly onset or chronic epilepsy and hoping to find whether there exist an autoimmune cause. whether the patients receive immune therapy or not will depend on the type and titter of the autoimmune antibody as well as the severity of the symptom. At 3 and 6 months later, all patients will be followed-up, and the positive autoimmune antibody will be redetected. the clinical manifest, clinical data, medication and treatment outcome will be recorded and analyzed, to study the diagnostic value of autoimmune antibody detection in new and chronic epilepsy

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with epilepsy according to the diagnostic criteria of International League Against Epilepsy (ILAE) 2017
* Age from 16 to 70 years old
* The etiology of patients with epilepsy is unknown
* The patient or guardian signs an informed consent and can cooperate with the inspection and follow-up for six months

Exclusion Criteria:

* Patients with hereditary, infectious, and metabolic epilepsy
* The investigation and follow-up cannot be completed due to vision, hearing, language expression, disturbance of consciousness, and impaired understanding, and the guardian cannot replace the completed
* Patients with other progressive or systemic diseases

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with newly onset or chronic epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
change of the seizure frequency | at six months after the patients being enrolled
  Seizure frequency are described as no seizures, less than one per month, monthly, weekly, and daily. the change of seizure frequency include 'increased', 'decreased', and 'no change' compared to the frequency before they were enrolled
change of the autoimmune antigen | at six months after the patients being enrolled
  autoimmune antigen in the serum of patients was described as positive and negative. the change of the autoimmune antigen include 'turn negative' and 'still positive' compared to the first detection.

IPD SHARING:
Plan to Share IPD: No